CLINICAL TRIAL: NCT02912325
Title: A Pilot, Non-Comparative Study to Assess the Efficacy and Safety of the New Food Supplement FaseMETS in Metabolic Syndrome
Brief Title: Non-Comparative Study to Assess the Efficacy and Safety of the New Food Supplement FaseMETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MDM S.p.A. (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPMDM/0216/FS
Record Dates: First submitted 2016-09-12; First posted 2016-09-23 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FaseMetS ® a food supplement (Other): Daily administration: 2 tablets FaseMETS a day
  Interventions: Dietary Supplement: Daily administration: 2 tablets FaseMETS a day

INTERVENTIONS:
Dietary Supplement: Daily administration: 2 tablets FaseMETS a day — Treatment with FaseMETS for 6 consecutive months in lowering serum lipids and glucose in subjects with Metabolic Syndrome

SUMMARY:
The primary objective is to evaluate the efficacy of FaseMETS for 6 consecutive months in lowering serum lipids and glucose in subjects with Metabolic Syndrome;

The secondary objectives of the trial are:

* to evaluate the potential benefit after 3 months of therapy (by an interim analysis)
* to evaluate the safety of FaseMETS

DETAILED DESCRIPTION:
The trial is designed as a multicenter, open label, non-comparative, 6 months, pilot study.

The primary objective is to evaluate the efficacy of FaseMetS ® administered for 6 months treatment combined with a health management plan in reducing the serum lipidemic profile (this includes total cholesterol, LDL cholesterol, HDL cholesterol, small density LDL particles, triglycerides, serum glucose, glycated haemoglobin (HBA1c), insulin, and pro-insulin, HOMA index, uric acid, body mass index (BMI), creatine phosphokinase) in patients diagnosed with Metabolic Syndrome and with mild to moderate Hypercholesterolemia.

The secondary objectives are:

* to evaluate the efficacy in reducing the serum lipidemic profile after a period of 3 months of FaseMetS ® ® treatment;
* to evaluate the safety of FaseMetS ® treatment by recording AE/SAE (with particular regards for gastrointestinal symptoms);
* improvement of blood clinical laboratory parameters;
* improvement of weight control systolic blood pressure and diastolic blood pressure control

ELIGIBILITY:
Inclusion Criteria:

* men or women
* age > 45 and ≤75 years
* on cardiovascular disease prevention in clinical practice
* written informed consent.
* total cholesterol≥200 mg/dL
* diagnosis of metabolic syndrome with three or more of the following:

  * Waist circumference: ≥89 cm for women and ≥102 cm for men or BMI≥25 Kg/m2;
  * Triglycerides level: ≥ 175 mg/dL or 1.7 mmol/L
  * HDL <40 mg/dL (1.04 mmol/L) in men or <50 mg/dL (1.3 mmol/L) in women
  * Blood sugar (fasting plasma glucose): ≥120 mg/dL (6.7 mmol/L)
  * Elevated blood pressure: systolic ≥ 130 and/or diastolic ≥ 85 mm Hg (antihypertensive drug treatment in a patient with a history of hypertension is an alternate indicator).

Exclusion Criteria:

* Pregnancy or lactation;
* Patients at very high or low cardiovascular risk, having a calculated SCORE ≥10% or <1% respectively
* History of atrial fibrillation or atrial flutter
* Patient in treatment with indication to oral anticoagulants or other antithrombotic drugs
* Patients with severe gastro-intestinal tract disorders with possible influence on drug absorption or electrolytes.
* Patients with myeloproliferative disorders
* Patients with severe chronic kidney disease (GFR 30 mL/min/ 1.73 m2), using Cockcroft's formula, with known liver disease or biliary obstructive disorders, chronic hepatitis, cirrhosis, with hyperkalemia or with ALAT or ASAT upper than 3 times the upper limit of normal laboratory range.
* History of alcoholism or drug abuse.
* Uncontrolled dysthyroidism, Cushing's syndrome, acromegalia, hyperparathyroidism.
* Patients with HIV or taking drugs for HIV.
* Patients taking statins or other dyslipidemic /hypolipidemic agents (drugs, food supplements, etc).
* Patients taking antidiabetic drugs (i.e metformin, acarbose and/or others).
* Patients unlikely to co-operate in the study or to comply well with treatment or with the study visits.
* Participation in another study at the same time or within the preceding 30 days.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Serum lipidemic profile evaluated at 6 months | 6 months
  laboratory test

SECONDARY OUTCOMES:
Serum lipidemic profile evaluated at 3 months | 3 months
  laboratory test
AE/SAE (with particular regards for gastrointestinal symptoms) | 6 months
  * blood clinical laboratory parameters
  * physical examination including weight, systolic blood pressure and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Maggi, MD, Study Director — MDM SpA Italy
Locations (2):
- Romania (2):
  - Opera Contract Research Organization SRL, Timișoara, Timiș County
  - Scm Dr Rosu, Timișoara, Timiș County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gielen S, Sandri M, Schuler G, Teupser D. Risk factor management: antiatherogenic therapies. Eur J Cardiovasc Prev Rehabil. 2009 Aug;16 Suppl 2:S29-36. doi: 10.1097/01.hjr.0000359233.58023.64. PMID 19675434
- [Background] Lorenzo C, Wagenknecht LE, D'Agostino RB Jr, Rewers MJ, Karter AJ, Haffner SM. Insulin resistance, beta-cell dysfunction, and conversion to type 2 diabetes in a multiethnic population: the Insulin Resistance Atherosclerosis Study. Diabetes Care. 2010 Jan;33(1):67-72. doi: 10.2337/dc09-1115. Epub 2009 Oct 6. PMID 19808919
- [Background] Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R; Cholesterol Treatment Trialists' (CTT) Collaborators. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. Lancet. 2005 Oct 8;366(9493):1267-78. doi: 10.1016/S0140-6736(05)67394-1. Epub 2005 Sep 27. PMID 16214597
- [Background] Cannon CP, Steinberg BA, Murphy SA, Mega JL, Braunwald E. Meta-analysis of cardiovascular outcomes trials comparing intensive versus moderate statin therapy. J Am Coll Cardiol. 2006 Aug 1;48(3):438-45. doi: 10.1016/j.jacc.2006.04.070. Epub 2006 Jul 12. PMID 16875966
- [Background] Alsheikh-Ali AA, Karas RH. The relationship of statins to rhabdomyolysis, malignancy, and hepatic toxicity: evidence from clinical trials. Curr Atheroscler Rep. 2009 Mar;11(2):100-4. doi: 10.1007/s11883-009-0016-8. PMID 19228482
- [Background] Joy TR, Hegele RA. Narrative review: statin-related myopathy. Ann Intern Med. 2009 Jun 16;150(12):858-68. doi: 10.7326/0003-4819-150-12-200906160-00009. PMID 19528564
- [Background] Rondanelli M, Giacosa A, Orsini F, Opizzi A, Villani S. Appetite control and glycaemia reduction in overweight subjects treated with a combination of two highly standardized extracts from Phaseolus vulgaris and Cynara scolymus. Phytother Res. 2011 Sep;25(9):1275-82. doi: 10.1002/ptr.3425. Epub 2011 Feb 10. PMID 21308825
- [Background] Luzzi R, Belcaro G, Hu S, Dugall M, Hosoi M, Ippolito E, Corsi M, Gizzi G. Beanblock(R) (standardized dry extract of Phaseolus vulgaris) in mildly overweight subjects: a pilot study. Eur Rev Med Pharmacol Sci. 2014 Oct;18(20):3120-5. PMID 25392114
- [Background] Bunnoy A, Saenphet K, Lumyong S, Saenphet S, Chomdej S. Monascus purpureus-fermented Thai glutinous rice reduces blood and hepatic cholesterol and hepatic steatosis concentrations in diet-induced hypercholesterolemic rats. BMC Complement Altern Med. 2015 Mar 28;15:88. doi: 10.1186/s12906-015-0624-5. PMID 25880551
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Oh HG, Kang YR, Lee HY, Kim JH, Shin EH, Lee BG, Park SH, Moon DI, Kim OJ, Lee IA, Choi J, Lee JE, Park KH, Suh JW. Ameliorative effects of Monascus pilosus-fermented black soybean (Glycine max L. Merrill) on high-fat diet-induced obesity. J Med Food. 2014 Sep;17(9):972-8. doi: 10.1089/jmf.2012.2740. Epub 2014 Aug 12. PMID 25115132
- [Background] Cicero AF, Morbini M, Rosticci M, D''Addato S, Grandi E, Borghi C. Middle-Term Dietary Supplementation with Red Yeast Rice Plus Coenzyme Q10 Improves Lipid Pattern, Endothelial Reactivity and Arterial Stiffness in Moderately Hypercholesterolemic Subjects. Ann Nutr Metab. 2016;68(3):213-9. doi: 10.1159/000445359. Epub 2016 Apr 8. PMID 27055107
- [Background] Patel S. Functional food red yeast rice (RYR) for metabolic syndrome amelioration: a review on pros and cons. World J Microbiol Biotechnol. 2016 May;32(5):87. doi: 10.1007/s11274-016-2035-2. Epub 2016 Apr 2. PMID 27038957
- [Background] McCarty MF, O'Keefe JH, DiNicolantonio JJ. Red Yeast Rice Plus Berberine: Practical Strategy for Promoting Vascular and Metabolic Health. Altern Ther Health Med. 2015;21 Suppl 2:40-5. PMID 26308759
- [Background] Burke FM. Red yeast rice for the treatment of dyslipidemia. Curr Atheroscler Rep. 2015 Apr;17(4):495. doi: 10.1007/s11883-015-0495-8. PMID 25728312
- [Background] Bhatnagar D, Soran H, Durrington PN. Hypercholesterolaemia and its management. BMJ. 2008 Aug 21;337:a993. doi: 10.1136/bmj.a993. No abstract available. PMID 18719012
- [Background] Brown P, Brunnhuber K, Chalkidou K, Chalmers I, Clarke M, Fenton M, Forbes C, Glanville J, Hicks NJ, Moody J, Twaddle S, Timimi H, Young P. How to formulate research recommendations. BMJ. 2006 Oct 14;333(7572):804-6. doi: 10.1136/bmj.38987.492014.94. PMID 17038740
- [Background] Connelly LM. Pilot studies. Medsurg Nurs. 2008 Dec;17(6):411-2. No abstract available. PMID 19248407